CLINICAL TRIAL: NCT04063969
Title: Analysis of the Radiation Safety Climate in the Hybrid Angiography Suite and Its Effects on Radiation Safety Performance
Brief Title: Analysis of the Radiation Safety Climate in the Hybrid Angiography Suite
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); AZ Sint-Jan AV (Other); Jan Yperman Ziekenhuis (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201837824
Record Dates: First submitted 2019-08-14; First posted 2019-08-21 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers; Aortic Aneurysm, Abdominal
Keywords: Radiation safety; Radiation safety climate; Radiation safety behavior; Quality improvement; Patient safety
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular team members: All vascular surgeons, surgical trainees, nurses active in the hybrid angiography suite at one of the participating centers will be invited to participate in the study.
  All participating team members complete an online questionnaire containing an assessment of their perceived radiation safety climate (28 items, 5 dimensions), radiation safety behaviors(2 items, 2 dimensions), radiation safety knowledge (single item) and radiation safety motivation (single item). All data will be stored pseudonymized.
  Interventions: Other: Assessment of radiation safety climate; Other: Assessment of radiation safety behavior; Other: Assessment of radiation safety knowledge and motivation
- Vascular surgical patients: In each center, five patients undergoing primary elective endovascular repair for an infrarenal abdominal aortic aneurysm (EVAR) will be enrolled in the study.
  For each participating patient, a set of demographical (BMI, case difficulty, ASA-grade,etc.), procedure-related (procedure duration, contrast use, etc.) and radiation dose parameters (DAP, cumulative air kerma) will be collected and stored in a pseudonymized way.
  Participation in this study has no effect on the interventional procedure, or the chosen approach.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Assessment of radiation safety climate — The rating tool contains 28 statements which cover 5 dimensions (Leadership, communication, commitment, resources, risk awareness) of the radiation safety climate. Participants are asked to indicate on a scale of 1 (completely disagree) - 3 (neutral) - 5 (completely agree) whether they agree with each statement. A composite radiation safety climate score is calculated by adding ratings on all items.
  Minimum scale score 28 - Maximum scale score 140
  Other Names: Radiation safety climate rating tool
  Groups: Endovascular team members
Other: Assessment of radiation safety behavior — The rating tool contains 2 statements which cover 2 dimensions of the radiation safety behavior. Participants are asked to indicate on a scale of 1 (completely disagree) - 3 (neutral) - 5 (completely agree) whether they agree with each statement. A composite radiation safety behavior score is calculated by adding ratings on both items Minimum scale score 2 - Maximum scale score 10
  Other Names: Radiation safety behavior rating tool
  Groups: Endovascular team members
Other: Assessment of radiation safety knowledge and motivation — The rating tool contains 2 statements which cover the radiation safety knowledge and behavior. Participants are asked to indicate on a scale of 1 (completely disagree) - 3 (neutral) - 5 (completely agree) whether they agree with each statement.
  Minimum item score 1 - maximum item score 5
  Other Names: Radiation safety knowledge and motivation rating tool
  Groups: Endovascular team members
Other: Data collection — Collection of patient-related data points Demographic information: ASA-classification, BMI Procedure related information: Procedural time, approach, contrast usage case difficulty Radiation safety parameters: Air Kerma, DAP, fluoroscopy time
  Groups: Vascular surgical patients

SUMMARY:
This study aims to measure the radiation safety climate in the hybrid angiography suite using self-assessment and to investigate the relationship of radiation safety climate with their self-reported safety behaviors.

The hypothesis is that a radiation safety climate does exist and can be measured using self-assessment. Additionally, it is expected that the radiation safety climate positively influences radiation safety behaviors.

DETAILED DESCRIPTION:
Radiation safety in the hybrid angiography suite is a primordial safety component which is relevant for endovascular team members and patients. To date, many interventions which aim to improve radiation safety habits of an endovascular team focus on improving technology and team radiation safety knowledge. Safety literature has indicated that a safety climate can be identified as the shared perceptions of team members or workers about the safety in their workspace and that this safety climate is closely related to safety behaviors and outcomes. In endovascular specialties, the concept of a radiation safety climate remains unexplored. Therefore, this study aims to measure the radiation safety climate in a diverse pool of endovascular team members from different hospitals, using self-assessment questionnaires and to investigate the relationship of radiation safety climate with their self-reported safety behaviors.

ELIGIBILITY:
Endovascular team member group

Inclusion Criteria:

* Vascular surgeon OR surgical trainee OR operating nurse
* Active at one of the participating hospitals

Exclusion Criteria:

* No exclusion criteria apply to this study.

Patient group Inclusion Criteria

* Patient undergoing elective endovascular repair of infrarenal abdominal aortic aneurysm

Exclusion criteria

* Emergency repair (ruptured aneurysm)
* Additional interventional procedures (iliac aneurysm, treatment of peripheral vessel disease)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Endovascular team members: vascular surgeons, surgical trainees, operating nurses
  * Patients undergoing elective endovascular repair of infrarenal abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Self-assessed radiation safety climate | Baseline measurement on study inclusion (Day 1)
  Radiation safety climate using radiation safety climate tool
Self-assessed radiation safety behavior | Baseline measurement on study inclusion (Day 1)
  Radiation safety behavior using radiation safety behavior tool
Self-assessed radiation safety knowledge and motivation | Baseline measurement on study inclusion (Day 1)
  Radiation safety knowledge and motivation using rating tool

SECONDARY OUTCOMES:
Procedural radiation doses - Dose area product | Registration during endovascular EVAR procedure - Within 1 week after patient study inclusion
  Procedural dose area product (DAP)
Procedural radiation doses - cumulative air kerma | Registration during endovascular EVAR procedure - Within 1 week after patient study inclusion
  Procedural cumulative air kerma (CAK)
Procedural radiation doses - fluoroscopy time | Registration during endovascular EVAR procedure - Within 1 week after patient study inclusion
  Procedural fluoroscopy time

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, MD, PhD, Principal Investigator — Vascular surgeon
Locations (5):
- Belgium (5):
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost Vlaanderen
  - Ghent University Hospital, Ghent, Oost Vlaanderen
  - AZ Sint Jan Brugge, Bruges, West Vlaanderen
  - Jan Yperman Ziekenhuis, Ieper, West Vlaanderen
  - GZA Campus Sint Augustinus, Antwerp

IPD SHARING:
Plan to Share IPD: No
Research data will not be shared standard

REFERENCES:
- [Background] Griffin MA, Neal A. Perceptions of safety at work: a framework for linking safety climate to safety performance, knowledge, and motivation. J Occup Health Psychol. 2000 Jul;5(3):347-58. doi: 10.1037//1076-8998.5.3.347. PMID 10912498